CLINICAL TRIAL: NCT04979208
Title: Impact of Changes in the Use of Care and Reorganization of the Healthcare System Linked to the Covid-19 Outbreak on the Quality of Care Pathways of Patients Suffering From Acute Myocardial Infarction and Stroke in the Aquitaine Region
Brief Title: Impact of Changes in the Use of Care and Reorganization of the Healthcare System Linked to the Covid-19 Outbreak on the Quality of Care Pathways of Patients Suffering From Acute Myocardial Infarction and Stroke in Aquitaine (AVICOVID)
Acronym: AVICOVID
Status: Completed | Type: Observational
Sponsor: University Hospital, Bordeaux (Other)
Responsible Party: Sponsor
Other Study IDs: CHUBX 2020/39
Record Dates: First submitted 2021-07-22; First posted 2021-07-28 (Actual); Last update posted 2021-08-11 (Actual); Status verified 2021-08

CONDITIONS: Coronavirus Disease 2019; Stroke; Acute Myocardial Infarction
Keywords: Stroke; Acute Myocardial Infarction; Coronavirus Disease 2019; Health Organization; Health Inequalities; Healthcare pathway
MeSH Terms: conditions — COVID-19; Stroke

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Acute myocardial infarction (AMI) cohort: Adult patients with recent acute myocardial infarction admitted to an hospital in the French Aquitaine region between January 1st 2019 and August 31 2020 and included in the ongoing, permanent, multicenter, retrospective and nominative ObA2 and REANIM/ACIRA registries. Were included in the analysis all recent AMI patients less than 24 hours old diagnosed by emergency physicians on the basis of suggestive clinical symptoms and electrocardiogram (ECG) criteria, cared in the 30 emergency units and 19 mobil intensive care unit, with a coronary angiography or a percutaneous coronary intervention (PCI) realized in the 11 cathlabs in Aquitaine
- Stroke cohort: Adult patients with recent stroke admitted to an hospital in the French Aquitaine region between January 1st 2019 and August 31 2020 and included in the ongoing, permanent, multicenter, retrospective and nominative ObA2 and REANIM/ACIRA registries. Were included in the analysis recent ischemic or hemorragic stroke patients with brain imaging managed in one of the 14 participating hospitals in Aquitaine (7 stroke units and 7 primary care centers).

SUMMARY:
The Covid-19 pandemic and its health and societal consequences raise fears of a deterioration in the management of non-Covid-19 pathologies, particularly those requiring rapid treatment. These fears relate in particular to strokes and acute myocardial infarctions (AMI), the two most frequent diseases, for which emergency treatment is a major factor in the vital and functional prognosis of patients. They are based on activity data from the emergency services, which have shown a sharp drop in admissions for AMI and strokes at the start of the pandemic. This drop is interpreted as being partly linked to a tendency for patients to delay or even give up care, which may be explained by fear of contamination, the desire not to solicit already overworked healthcare professionals and overload in emergency structures. In addition, studies have shown that the time required to treat AMI during the pandemic phase in China has been extended due to the new organizations set up in healthcare institutions in connection with this major health event. In addition, certain inequalities in access to care, already identified during the non- pandemic period among AMI and stroke patients, are likely to be accentuated by the new healthcare organizations set up during the pandemic period.

The investigators are interested in the impact of changes in healthcare utilization and reorganization within hospitals, related to the Covid-19 pandemic, on the quality of the care pathway for stroke and AMI patients in the Aquitaine region. The investigators also study the role of the socio-demographic, socio-economic and geographical characteristics of these patients as factors of inequality of access to care during this period.

The project is based on data collected within the Aquitaine Cardio-Neuro-Vascular Registries (CNV), an exhaustive cohort of stroke and AMI patients treated by a health care institution in Aquitaine. They are an excellent tool for describing the care pathway and outcomes of these patients, from the onset of symptoms to the end of the acute episode. An additional collection is planned to collect all the organizations and activities set up within the hospitals in Aquitaine. The study period, from January 2019 to August 2020, provides sufficient time before lockdown and after the date of the end of lockdown, to analyze trends in the quality of pathways, according to the various reorganizations of the health system and changes in the use of care linked to the management of the Covid-19 pandemic.

The project identifies the reorganizations with the most striking consequences on the quality of care for patients suffering from non Covid-19 pathologies. It analyzes the changes in the behaviour of patients and their family and caregivers in their use of care during the Covid-19 pandemic and their impact on the care pathways and results. It contributes to the policy of reducing inequalities in access to care and to the definition of a health strategy in the event of a major health crisis.

ELIGIBILITY:
Inclusion Criteria:

* Patients over 18 years, domiciled in metropolitan France
* Patients managed between January 1st 2019 and August 31 2020, by emergency units in Aquitaine for AMI
* Patients managed between January 1st 2019 and August 31 2020, by emergency units in Aquitaine for recent stroke

Exclusion Criteria:

AMI cohort :

* Patient with pacemaker;
* Patients in cardiac arrest before performing the first qualifying ECG.

Stroke cohort :

- Patients treated for sequelae rehabilitation, complications of a recent stroke, transient ischemic accident or any other neurological pathology

Both :

Patients who refused to participate

Min Age: 18 Years | Sex: All
Age Groups: Adult, Older Adult
Study Population: Patients managed between January 1st 2019 and August 31 2020, by emergency units in Aquitaine for an AMI or a recent stroke
Sampling Method: Non-Probability Sample
Enrollment: 9218 (Actual)
Dates: Start 2020-07-15 (Actual); Primary Completion 2021-07-09 (Actual); Study Completion 2021-07-09 (Actual)

PRIMARY OUTCOMES:
Delay for AMI patient | At inclusion in the cohort during the acute episode
  Delay between the first medical contact and the procedure (coronary angiography or Percutaneous Coronary Intervention)
Delay for stroke patient | At inclusion in the cohort during the acute episode
  Delay between the admission to hospital and the imagery

CONTACTS AND LOCATIONS:
Locations (1):
- CHU Bordeaux, Bordeaux, France

REFERENCES:
- [Derived] Lesaine E, Francis F, Domecq S, Miganeh-Hadi S, Sevin F, Sibon I, Rouanet F, Pradeau C, Coste P, Cetran L, Vandentorren S, Saillour F; AVICOVID group. Social and clinical vulnerability in stroke and STEMI management during the COVID-19 pandemic: a registry-based study. BMJ Open. 2024 Jan 3;14(1):e073933. doi: 10.1136/bmjopen-2023-073933. PMID 38171619
- [Derived] Lesaine E, Francis-Oliviero F, Domecq S, Bijon M, Cetran L, Coste P, Lhuaire Q, Miganeh-Hadi S, Pradeau C, Rouanet F, Sevin F, Sibon I, Saillour-Glenisson F; AVICOVID group. Effects of healthcare system transformations spurred by the COVID-19 pandemic on management of stroke and STEMI: a registry-based cohort study in France. BMJ Open. 2022 Sep 21;12(9):e061025. doi: 10.1136/bmjopen-2022-061025. PMID 36130741
- See also: Related Info — https://www.registres-cnv.fr/